CLINICAL TRIAL: NCT03130296
Title: Genotyping FcɣRs Genes of HIV-1 Patients "Progressor": Correlation With the Changing Profile of the Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6493
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: HIV Infection
Keywords: HIV infection; Fc receptor polymorphism (FcR)
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This non-interventional study aims to determine whether there is a correlation between the Fc receptor polymorphism (FcR) and the course of the disease following HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or older,
* Patient affiliated to a social security scheme,
* Informed consent dated and signed by the investigating physician the patient,
* Patients infected with HIV-1 having progressed in clinical (stage C) or biologically (CD4 nadir <350 / mm3 and viral load> 10,000 copies / ml)

Exclusion Criteria:

* Impossibility of giving the subject informed information (subject in an emergency situation, difficulty in understanding the subject, ...)
* Subject under safeguard of justice,
* Subject under tutelage or under curatorship,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with HIV-1 having progressed in clinical (stage C) or biologically (CD4 nadir <350 / mm3 and viral load> 10,000 copies / ml)
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-02-16 (Estimated); Study Completion 2020-02-16 (Estimated)

PRIMARY OUTCOMES:
Correlation research between Fc receptor polymorphism (FcR) and the course of disease following HIV infection. | After infection, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David REY, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Le Trait d'Union - Centre de soins de l'infection par le VIH au NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No